CLINICAL TRIAL: NCT04590859
Title: Penile Blood Flow Characteristics Following Caudal or Penile Block
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Adam Adler MD, MS, FAAP, Assistant Professor, Baylor College of Medicine
Other Study IDs: H-48138
Record Dates: First submitted 2020-09-10; First posted 2020-10-19 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: The Aim of This Study is to Measure Blood Flow Before and After a Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Penile block: Patients undergoing procedure with penile block
  Interventions: Procedure: Block performed; Device: LMA placement
- caudal block: Patients undergoing procedure with caudal block
  Interventions: Procedure: Block performed; Device: LMA placement

INTERVENTIONS:
Procedure: Block performed — Comparing block performed with penile blood flow
Device: LMA placement — Placement of LMA for airway securement

SUMMARY:
Pediatric urologic surgery is generally accompanied by use of a caudal or penile block for analgesia. A caudal block is performed by injecting local anesthetic in the low epidural space while a penile block is performed by injecting local anesthetic above the pubic symphysis. Local anesthetic in the epidural space is known to caudal vasodilation interiorly. It is unknown as to whether this vasodilation results in alteration in flow to the penile tissue and potentially changes tissue characteristics. The aim of this study is to measure blood ultrasound velocity in the dorsal penile artery and vein before and after a block.

DETAILED DESCRIPTION:
Pediatric urologic surgery is generally accompanied by use of a caudal or penile block for analgesia. A caudal block is performed by injecting local anesthetic in the low epidural space while a penile block is performed by injecting local anesthetic above the pubic symphysis. Local anesthetic in the epidural space is known to caudal vasodilation interiorly. It is unknown as to whether this vasodilation results in alteration in flow to the penile tissue and potentially changes tissue characteristics. The aim of this study is to measure blood ultrasound velocity in the dorsal penile artery and vein before and after a block.

ELIGIBILITY:
Inclusion Criteria:

* Children ages <7 years undergoing circumcision at TCH Penile or Caudal block to be performed at discretion of anesthesiology/Urology providers
* ASA classification1,2
* use of laryngeal mask airway

Exclusion Criteria:

* Previous cardiac surgery
* Antihypertensive medication
* requirement for intravenous anesthetic
* ASA classification non 1,2
* parental refusal of participation parental refusal of block
* patients requiring intubation

Ages: 2 Years to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — penile study only applicable to males
Study Population: males undergoing circumcision using penile or caudal
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
penile blood flow | 20 minutes
  assessment of changes using ultrasound to blood flow based on block performed

CONTACTS AND LOCATIONS:
Locations (1):
- Texas childrens Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided